CLINICAL TRIAL: NCT04328987
Title: Safety of Cold Snare Polypectomy in Patients With Uninterrupted Antiplatelet Agent : Aspirin vs Clopidogrel
Brief Title: Safety of Cold Snare Polypectomy in Patients With Uninterrupted Antiplatelet Agent
Status: Completed | Type: Observational
Sponsor: Incheon St.Mary's Hospital (Other)
Collaborators: Seoul St. Mary's Hospital (Other); St Vincent's Hospital (Other); Uijeongbu St. Mary's Hospital (Unknown); Soonchunhyang University Hospital (Other); Bucheon St. Mary's Hospital (Other); Eunpyeong St. Mary's Hospital (Other); Gangneung Asan Hospital (Other); Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Geun Gweon, Assistant Professor, Incheon St.Mary's Hospital
Other Study IDs: XC19OCDI0089
Record Dates: First submitted 2020-03-28; First posted 2020-04-01 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Post Polypectomy Bleeding
Keywords: antiplatelet agent; aspirin; clopidogrel; cold snare polypectomy; safety; post polypectomy bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Clopidogrel user: * Uninterrupted (continuous) use of clopidogrel: cessation of clopidogrel less than 4 days (=0, 1, 2, or 3 days cessation). Cessation days of clopidogrel is sum of before and after the CSP
  1. patient who stopped clopidogrel only on the day of colonoscopy and resumed the day after colonoscopy -> cessation of clopidogrel was 1 day.
  2. patient who stopped clopidogrel from 3 days before colonoscopy and resumed the day after colonoscopy -> cessation of clopidogrel was 4 days (-3, -2, -1, 0=on the day of colonoscopy). -> interruption of clopidogrel -> excluded from study.
  3. patient who stopped clopidogrel from 2 days before colonoscopy and resumed 2 days after colonoscopy -> cessation of clopidogrel was 4 days (-2, -1, 0=on the day of colonoscopy, 1=the day after colonoscopy). -> interruption of clopidogrel -> excluded from study.
  Interventions: Procedure: cold snare polypectomy
- Aspirin user: * Uninterrupted (continuous) use of aspirin: cessation of aspirin less than 4 days (=0, 1, 2, or 3 days cessation). Cessation days of aspirin is sum of before and after the CSP
  1. patient who stopped aspirin only on the day of colonoscopy and resumed the day after colonoscopy -> cessation of aspirin was 1 day.
  2. patient who stopped aspirin from 3 days before colonoscopy and resumed the day after colonoscopy -> cessation of aspirin was 4 days (-3, -2, -1, 0=on the day of colonoscopy). -> interruption of aspirin -> excluded from study.
  3. patient who stopped aspirin from 2 days before colonoscopy and resumed 2 days after colonoscopy -> cessation of aspirin was 4 days (-2, -1, 0=on the day of colonoscopy, 1=the day after colonoscopy). -> interruption of aspirin -> excluded from study.
  Interventions: Procedure: cold snare polypectomy

INTERVENTIONS:
Procedure: cold snare polypectomy — Resection of colorectal polyp using cold snare polypectomy method. The polyp will be resected by mechanical force of snare without electrical cautery.

SUMMARY:
Polypectomy is regarded as high risk for bleeding. Several guidelines recommend continuous use of aspirin during polypectomy. However for clopidogrel, widely used antiplatelet agent, cessation of 5-7 is recommended. There is insufficient data regarding clopidogrel on post polypectomy bleeding. Delayed bleeding after polypectomy in patients with clopidogrel was reported as 3%. A recent study showed that delayed bleeding rate in patients with clopidogrel didn't differ that of who stopped clopidogrel. However the rate for delayed bleeding was 4%, higher than the previous studies. More studies are needed to conclude the safety of polypectomy in clopidogrel users.

Cold snare polypectomy (CSP) can resect polyps without electrical energy. CSP are safe than conventional endoscopic mucosal resection in high risk for bleeding.

The polypectomy techniques in most of studies were heterogenous, where delayed bleeding was investigated in clopidogrel users. There is no study to investigate safety of CSP in patients with clopidogrel users to date. The investigators hypothesized that the bleeding risk of CSP in patients with clopidogrel users would be similar to that of aspirin users.

In this multicenter prospective study, the investigators aimed to compare the safety of CSP between aspirin and clopidogrel users.

DETAILED DESCRIPTION:
* Cold snare polypectomy (CSP): resection of colorectal polyp by mechanical force of snare, without electric cautery.
* Antiplatelet agent: single use of aspirin or clopidogrel
* Uninterrupted (continuous) use of antiplatelet agent: cessation of antiplatelet agent less than 4 days. Cessation of antiplatelet agent is sum of before and after the CSP

ex.)

1. patient who stopped aspirin only on the day of colonoscopy and resumed the day after colonoscopy -> cessation of aspirin was 1 day.
2. patient who stopped aspirin only on the day of colonoscopy and resumed the 2 days after colonoscopy -> cessation of aspirin was 2 days (before colonoscopy 1day + after colonoscopy 1day).
3. patient who stopped aspirin from 3 days before colonoscopy and resumed the day after colonoscopy -> cessation of aspirin was 4 days (-3, -2, -1, 0=on the day of colonoscopy). -> interruption of aspirin -> excluded from study.
4. patient who stopped aspirin from 2 days before colonoscopy and resumed 2 days after colonoscopy -> cessation of aspirin was 4 days (-2, -1, 0=on the day of colonoscopy, 1=the day after colonoscopy). -> interruption of aspirin -> excluded from study.

   * BLEEDING # Immediate (intraprocedural) bleeding After CSP, bleeding will be observed for 2 minutes. Bleeding grade: (1) no bleeding, (2) minor (negligible) bleeding, (3) major bleeding, and (4) active bleeding (spurting).

In case of Grade 3 or 4, hemoclipping will be applied

* Delayed bleeding Delayed bleeding will be defined when all of the following criteria were met: (1) anal bleeding after discharge of endoscopy unit and (2) identification of polypectomy bleeding site by colonoscopy.
* Significant delayed bleeding Any of the following criteria: (1) hemoglobin drop >2, (2) hemodynamic instability, (3) admission, (4) transfusion, and (5) surgery or angiography for hemostasis.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-80
* polyp size <10mm
* polyp resection : cold snare polypectomy
* cessation of antiplatelet agent less than 4 days

Exclusion Criteria:

* ASA class IV or above,
* hematologic diseases including idiopathic thrombocytopenic purpura, leukemia, and aplastic anemia
* advanced liver cirrhosis
* cessation of antiplatelet agent for 4 days or more
* dual antiplatelet agent users
* coagulopathy (abnormal PT, aPTT, or platelet count)

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Uninterrupted (continuous) use of antiplatelet agent: cessation of antiplatelet agent less than 4 days. Cessation of antiplatelet agent is sum of before and after the CSP
  ex.)
  1. patient who stopped aspirin only on the day of colonoscopy and resumed the day after colonoscopy -> cessation of aspirin was 1 day.
     (before colonoscopy 1day + after colonoscopy 1day).
  2. patient who stopped aspirin from 2 days before colonoscopy and resumed 2 days after colonoscopy -> cessation of aspirin was 4 days (-2, -1, 0=on the day of colonoscopy, 1=the day after colonoscopy). -> interruption of aspirin -> excluded from study.
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Delayed post polypectomy bleeding | From discharge of endoscopy unit until 4 weeks after polypectomy
  Delayed bleeding will be defined when all of the following criteria were met: (1) anal bleeding after discharge of endoscopy unit and (2) identification of polypectomy bleeding site by colonoscopy.

SECONDARY OUTCOMES:
Immediate bleeding (intraprocedural bleeding) | until 2 minutes after polypectomy
  Bleeding 2 minutes after polypectomy.
  (1) no bleeding, (2) minor (negligible) bleeding, (3) major bleeding, and (4) active bleeding (spurting).

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Gun Kim, MD, Ph.D, Study Chair — Soonchunhyang University Hospital
Locations (1):
- Bucheon St. Mary's Hospital, Bucheon-si, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gweon TG, Kim HG, Jung Y, Jeon SR, Na SY, Lee YJ, Kim TH. Safety of cold snare resection techniques for removal of polyps in the small colon in patients taking clopidogrel and aspirin: a Korean Association for the Study of Intestinal Diseases prospective multicenter study. Gastrointest Endosc. 2025 Apr;101(4):866-876. doi: 10.1016/j.gie.2024.10.014. Epub 2024 Oct 16. PMID 39424007